CLINICAL TRIAL: NCT04164212
Title: Live Attenuated Influenza Vaccine as a Nasal Model for Influenza Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Lafon, Clinical Instructor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300004274; R01HL149944 (NIH)
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- open label (Other): FLUMIST QUADRIVALENT 0.2 mL dose supplied in a single-dose pre-filled intranasal sprayer
  Interventions: Drug: Flumist Quadrivalent Nasal Product

INTERVENTIONS:
Drug: Flumist Quadrivalent Nasal Product — FLUMIST QUADRIVALENT 0.2 mL dose supplied in a single-dose pre-filled intranasal sprayer
  Other Names: live attenuated influenza vaccine

SUMMARY:
The purpose of this study is to develop a nasal model for influenza infection using the live attenuated influenza vaccine (LAIV). The investigators will administer LAIV to healthy adult volunteers in order to simulate influenza infection, and obtain nasal specimens to measure influenza virus and inflammatory/immune responses. In a subset of participants, cystic fibrosis transmembrane conductance regulator (CFTR) function will also be evaluated via measurement of nasal potential difference (NPD)

ELIGIBILITY:
Inclusion Criteria:

* ages 18-49 years old,
* not yet received influenza vaccine for 2019-2020, and
* capable of giving signed informed consent.

Exclusion Criteria:

* Immunocompromising condition (e.g. HIV/AIDS, chemotherapy, immune suppressing medications),
* active smoking within past 6 months,
* asthma, chronic lung/liver/kidney /neurologic/hematologic/metabolic disorders,cardiovascular disease (excluding isolated hypertension), diabetes mellitus, disease, congestive heart failure,
* pregnancy,
* current or recent (within the past month) upper/lower respiratory tract infection, chronic sinusitis/nasal allergies requiring frequent or daily therapy (including topical corticosteroids),
* prior adverse reaction to influenza vaccine,
* history of Guillain-Barre syndrome,
* egg allergy,
* close contact with an individual with severe immunodeficiency/immunosuppression.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
influenza virus replication | day 2
  virus replication will be measured using RT-PCR and reported as genomic units, from samples obtained from nasal washing and nasal oropharyngeal swabs
markers of inflammation | change in inflammatory cytokines from baseline to day 2
  a standard panel of inflammatory cytokines (Luminex Performance Human XL Cytokine Discovery Panel assay, R&D Systems; results reported in pg/ml) will be measured in samples obtained from nasal washing and nasal oropharyngeal swabs
cystic fibrosis transmembrane conductance regulator function | change in NPD from baseline to day 2
  nasal potential difference (NPD) measurement

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States